CLINICAL TRIAL: NCT00740207
Title: A Phase IV Pilot Study to Compare ISOVUE®-250 and VISIPAQUE™ 270 for Motion Artifact and Pain in Peripheral Digital Subtraction Angiography (DSA)
Brief Title: Pilot Study to Compare ISOVUE®-250 and VISIPAQUE™ 270 for Motion Artifact and Pain in Peripheral DSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Carmela Houston/ Sr. Manager Corporate Clinical Research, Bracco Diagnostics
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IOP-113
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-05

CONDITIONS: Peripheral Arterial Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1 | interventions — iodixanol; Iopamidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Isovue 250 (Active Comparator)
  Interventions: Drug: Isovue 250
- VISIPAQUE 270 (Active Comparator)
  Interventions: Drug: VISIPAQUE 270

INTERVENTIONS:
Drug: VISIPAQUE 270 — VISIPAQUE 270 (Iodixanol Injection) is provided in bottles/flexible containers, ready to use sterile, pyrogen-free colorless to pale yellow solution
  Other Names: Iodixanol Injection
  Arms: VISIPAQUE 270
Drug: Isovue 250 — ISOVUE-250 (Iopamidol Injection) is provided in single dose bottles/vials, ready to use, aqueous, nonpyrogenic, colorless to pale yellow sterile solution
  Other Names: Iopamidol Injection
  Arms: Isovue 250

SUMMARY:
The purpose of this study is to compare ISOVUE-250 and VISIPAQUE 270 for motion artifact and pain following intraarterial injection for peripheral DSA.

ELIGIBILITY:
Inclusion Criteria:

Enroll a patient in this study if the patient meets the following inclusion criteria:

* Provides written Informed Consent and is willing to comply with protocol requirements;
* Is at least 18 years of age;
* Is scheduled to undergo peripheral DSA for the diagnosis and/or treatment (PTA) of PAOD.

Exclusion Criteria:

Exclude a patient from this study if the patient does not fulfill the inclusion criteria, or if any of the following conditions are observed:

* Is a pregnant or lactating female. Exclude the possibility of pregnancy:
* by testing on site at the institution (serum or urine βHCG) within 24 hours prior to the start of investigational product administration,
* by surgical history (e.g., tubal ligation or hysterectomy),
* post menopausal with a minimum 1 year without menses;
* Has any known allergy to one or more of the ingredients of the investigational products;
* Has a history of severe congestive heart failure [class IV in accordance with the classification of the New York Heart Association (NYHA)]
* Was previously entered into this study or received an investigational compound within 30 days before admission into this study;
* Has a history of hypersensitivity to iodinated contrast agents;
* Has renal impairment (eGFR <60 mL/min/1.73 m2, calculated using the Modification of Diet in Renal Disease [MDRD] study equation , );
* Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or postdose follow-up examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven N. Sireci, MD, Study Chair — Bracco Diagnostics, Inc

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first patient to participate in this study was dosed on September 17, 2008; the last patient on June 15, 2009.
Groups:
- ISOVUE 250; VISIPAQUE 270: Participants were injected at least once in 1 of the following 3 locations: aortic bifurcation (injection rate 8-10 mL/s, total volume 15-20 mL), iliac arteries (injection rate 5-6 mL/s, total volume 10-12 mL), or superficial femoral artery (injection rate 3-5 mL/s, depending on diameter and condition of artery, total volume 8-12 mL to view only thigh, 10-15 mL to view calf as well, 20 mL for full runoff to foot).
Period: Overall Study
Arm/Group | ISOVUE 250 | VISIPAQUE 270
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ISOVUE 250 | VISIPAQUE 270 | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 7 | 13
  >=65 years | 11 | 9 | 20
Age Continuous [Mean (Standard Deviation); unit: years] | 65.9 (9.42) | 66.9 (9.93) | 66.4 (9.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13
  Canada | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Level of Pain in the Lower Extremities Scored by the Participants on the Visual Analog Scale Following Intraarterial Administration of ISOVUE-250 or VISIPAQUE 270 in Peripheral DSA.
Description: Visual Analog Scale: Patients were asked to mark on a 10 centimeter line where their pain was in the lower extremity of interest, in relation to the 2 extremes: no pain (0) on the far left and worst pain (10) on the far right. Pain Severity Scale: (0) None = VAS Score 0; (1) Mild = VAS Score 1-3; (2) Moderate = VAS Score 4-6; (3) Severe = VAS Score 7-10. Patients were assessed immediately prior to injection and again immediately following injection.
Time Frame: Immediately prior to power injection run and again immediately following power injection run
Population: Patients who did not deviate from the planned protocol.
Measure: Number; unit: Participants
Groups:
- VAS Score Prior to Injection of ISOVUE 250; VAS Score Prior to Injection of VISIPAQUE 270: Pain Severity Scale: (0) None = VAS Score 0; (1) Mild = VAS Score 1-3; (2) Moderate = VAS Score 4-6; (3) Severe = VAS Score 7-10.
- VAS Score After Injection of ISOVUE 250; VAS Score After Injection of VISIPAQUE 270: Participants were injected at least once in 1 of the following 3 locations: aortic bifurcation (injection rate 8-10 mL/s, total volume 15-20 mL), iliac arteries (injection rate 5-6 mL/s, total volume 10-12 mL), or superficial femoral artery (injection rate 3-5 mL/s, depending on diameter and condition of artery, total volume 8-12 mL to view only thigh, 10-15 mL to view calf as well, 20 mL for full runoff to foot).
Arm/Group | VAS Score Prior to Injection of ISOVUE 250 | VAS Score After Injection of ISOVUE 250 | VAS Score Prior to Injection of VISIPAQUE 270 | VAS Score After Injection of VISIPAQUE 270
Number analyzed (Participants) | 10 | 10 | 10 | 10
Participants
  (0) None | 8 (1.35) | 6 (1.03) | 7 | 2
  (1) Mild | 0 | 1 | 1 | 7
  (2) Moderate | 2 | 3 | 2 | 1
  (3) Severe | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: VAS Score After Injection of ISOVUE 250 vs VAS Score After Injection of VISIPAQUE 270; Paired t-test to compare difference between the investigational product's mean change from predose to postdose; Test type: Superiority or Other; p = 0.7142, t-test, 2 sided; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.3 to 0.9]

2. Secondary Outcome: The Number of Participants With Motion Artifacts Following Intraarterial Administration of ISOVUE-250 or VISIPAQUE 270 in Peripheral DSA.
Description: Using the following 5-point scale, the Investigator reviewed the images for motion artifact in vessels distal to the knee: 0 = None; 1 = Mild, not significant; 2 = Significant, but correctable; 3 = Degrades image quality; 4 = Images uninterpretable.
Time Frame: Immediately postdose
Population: Patients who did not deviate from the planned protocol.
Measure: Number; unit: Participants
Arm/Group | ISOVUE 250 | VISIPAQUE 270
Number analyzed (Participants) | 10 | 10
Participants
  (0) No Motion Artifacts | 8 | 4
  (1) Mild, Not significant | 1 | 5
  (2) Significant, But Correctable | 1 | 1
  (3) Degrades Image Quality | 0 | 0
  (4) Images Uninterpretable | 0 | 0
Statistical Analysis 1: Comparison: ISOVUE 250 vs VISIPAQUE 270; Paired t-test to compare the difference in percentage between the portions of patients who had motion artifacts; Test type: Superiority or Other; p = 0.1698, Fisher Exact; Mean Difference (Final Values) = -40.0, 95% CI 2-sided [-79.2 to -0.8]

3. Secondary Outcome: The Number of Participants Requiring Repeat Injection(s) Following Intraarterial Administration of ISOVUE-250 or VISIPAQUE 270 in Peripheral DSA.
Description: The Investigator assessed the images and recorded the number of repeat power injections required due to motion artifacts for each participant.
Time Frame: Immediately postdose
Measure: Number; unit: Participants
Arm/Group | ISOVUE 250 | VISIPAQUE 270
Number analyzed (Participants) | 10 | 10
Participants | 0 | 1
Statistical Analysis 1: Comparison: ISOVUE 250 vs VISIPAQUE 270; Paired t-test to compare difference in percentage between the number of participants requiring repeat injections; Test type: Superiority or Other; p = 1.000, Fisher Exact; Mean Difference (Final Values) = -10.0, 95% CI 2-sided [-28.6 to 8.6]

ADVERSE EVENTS:
Arm/Group | ISOVUE 250 | VISIPAQUE 270
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 1/17 | 0/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISOVUE 250 (N=17) | VISIPAQUE 270 (N=16)
Procedural Complication/Right Groin Bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be presented during scientific symposia or published in a scientific journal only after review by Bracco in accordance with the guidelines set forth in the applicable publication or financial agreement.